CLINICAL TRIAL: NCT03250832
Title: A Phase 1 Dose Escalation and Cohort Expansion Study of TSR-033, an Anti-LAG-3 Monoclonal Antibody, Alone and in Combination With an Anti-PD-1 in Patients With Advanced Solid Tumors
Brief Title: Study of TSR-033 With an Anti-programmed Cell Death-1 Receptor (PD-1) in Participants With Advanced Solid Tumors
Acronym: CITRINO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 213349; 4040-01-001 (Other: Tesaro)
Record Dates: First submitted 2017-06-22; First posted 2017-08-16 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Neoplasms
Keywords: Advanced solid tumors; Dostarlimab; Ovarian cancer; Colorectal cancer; Lung cancer; Dose escalation; Dose expansion
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms; Lung Neoplasms | interventions — TSR-033; dostarlimab; IFL protocol; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1a: TSR-033 monotherapy dose escalation (Experimental): Part 1a will evaluate TSR-033 at ascending doses (20 milligrams [mg], 80 mg and 240 mg) every 2 weeks. Cohorts will be enrolled sequentially and will initially follow a 3+3 design at a starting dose of 20 mg.
  Interventions: Drug: TSR-033
- Part 1b: TSR-033 monotherapy PK/PDy characterization (Experimental): Part 1b will evaluate the PK profile and assess PDy data from blood and tumor tissue samples following TSR-033 treatment. The participants will begin treatment with TSR-033 on Day 1 followed by 28 days observation for collection of blood sampling for PK/PDy. Participants will receive their second dose of TSR-033 on Day 29 and every 14 days thereafter.
  Interventions: Drug: TSR-033
- Part 1c: TSR-033+dostarlimab combination dose escalation (Experimental): Participants will be administered ascending doses of TSR-033 in combination with dostarlimab 500 mg every 3 weeks. Planned dose levels of TSR-033 include 80 and 240 mg.
  Interventions: Drug: TSR-033; Drug: Dostarlimab
- Part 2 Cohort A: TSR-033+dostarlimab combination (Experimental): Part 2 Cohort A will evaluate the preliminary activity of TSR-033 in combination with dostarlimab in anti-PD-1 naive participants with third and fourth line MSS-CRC. TSR-033 will be administered every 2 weeks and dostarlimab every 6 weeks.
  Interventions: Drug: TSR-033; Drug: Dostarlimab
- Part 2 Cohort B1: TSR-033+dostarlimab with mFOLFOX6 (Experimental): Part 2 Cohort B1 will evaluate the preliminary activity of TSR-033 administered every 2 weeks (Q2W) in combination with dostarlimab administered every 6 weeks (Q6W) along with mFOLFOX6 and bevacizumab (standard of care [SOC]) in anti-PD-1 naive second line MSS-CRC participants who have progressed on frontline treatment with FOLFIRI, with or without biologics.
  Interventions: Drug: TSR-033; Drug: Dostarlimab; Drug: mFOLFOX6; Drug: Bevacizumab
- Part 2 Cohort B2: TSR-033+dostarlimab with FOLFIRI (Experimental): Part 2 Cohort B2 will evaluate the preliminary activity of TSR-033 in combination with FOLFIRI and bevacizumab (SOC) in anti-PD-1 naive second line MSS-CRC participants who have progressed on frontline treatment with FOLFOX, with or without biologics.
  Interventions: Drug: TSR-033; Drug: Dostarlimab; Drug: FOLFIRI; Drug: Bevacizumab

INTERVENTIONS:
Drug: TSR-033 — TSR-033 is a humanized monoclonal antibody immunoglobulin (Ig) G4.
  Other Names: LAG-3
Drug: Dostarlimab — Dostarlimab (previously referred to as TSR-042) is an IgG4 antibody.
  Arms: Part 1c: TSR-033+dostarlimab combination dose escalation; Part 2 Cohort A: TSR-033+dostarlimab combination; Part 2 Cohort B1: TSR-033+dostarlimab with mFOLFOX6; Part 2 Cohort B2: TSR-033+dostarlimab with FOLFIRI
Drug: mFOLFOX6 — mFOLFOX6 is combination of folinic acid (FOL)/leucovorin, 5-fluorouracil and oxaliplatin (OX) which acts as systemic cytotoxic agent.
  Arms: Part 2 Cohort B1: TSR-033+dostarlimab with mFOLFOX6
Drug: FOLFIRI — FOLFIRI is combination of folinic acid (FOL)/leucovorin, 5-fluorouracil and irinotecan (IRI) which acts as systemic cytotoxic agent.
  Arms: Part 2 Cohort B2: TSR-033+dostarlimab with FOLFIRI
Drug: Bevacizumab — Bevacizumab is a humanized monoclonal IgG1 antibody that targets vascular endothelial growth factor (VEGF)-A to inhibit angiogenesis.
  Arms: Part 2 Cohort B1: TSR-033+dostarlimab with mFOLFOX6; Part 2 Cohort B2: TSR-033+dostarlimab with FOLFIRI

SUMMARY:
This is a multicenter, open-label, first-in-human Phase 1 study evaluating the anti-lymphocyte activation gene-3 (LAG-3) antibody TSR-033 alone, in combination with the anti-PD-1 antibody dostarlimab, and in combination with dostarlimab, modified folinic acid (FOL)/leucovorin, 5-fluorouracil and oxaliplatin (OX) (mFOLFOX6) or FOL/leucovorin, 5-fluorouracil and irinotecan (IRI) (FOLFIRI), and bevacizumab in participants with advanced solid tumors in a broad range of solid tumors. Participants with disease types selected for evaluation in this study are expected to derive clinical benefit with addition of an anti-PD-1. The study will be conducted in two parts with Part 1 consisting of dose escalation to determine the recommended phase 2 dose (RP2D) of TSR-033 as a single agent (Part 1a) and in combination with dostarlimab (Part 1c). RP2D decisions will be based on the occurrence of dose-limiting toxicities (DLTs), pharmacokinetics (PK), as well as pharmacodynamics (PDy) data. Part 2A of the study will investigate the anti-tumor activity of TSR-033 and dostarlimab in combination in participants with advanced or metastatic microsatellite stable colorectal cancer (MSS-CRC). Part 2B of the study will investigate the safety and anti-tumor activity of TSR-033 and dostarlimab in combination with chemotherapy (Cohort B1: mFOLFOX6 and Cohort B2: FOLFIRI) and bevacizumab in participants with advanced or metastatic MSS-CRC.

ELIGIBILITY:
Inclusion Criteria for participants in Part 1:

* The participant is >=18 years of age.
* The participant has any histologically or cytologically confirmed advanced (unresectable) or metastatic solid tumor and has PD after treatment with available therapies that are known to confer clinical benefit or who are intolerant to treatment.
* The participant must have an archival tumor tissue sample that is formalin-fixed and paraffin-embedded (FFPE) (blocks preferred over slides) and requested and confirmed available from offsite locations prior to dosing. The quality and quantity of the sample must be confirmed sufficient as per the Study Laboratory Manual. Participants who do not have archival tissue must agree to a new biopsy to obtain fresh tumor tissue prior to dosing.
* Part 1b (PK/PDy cohort): The participant must have lesions amenable for biopsy and agree to undergo biopsies for fresh tumor tissue prior to treatment, approximately 4 to 6 weeks after treatment, and, whenever possible, at the time of PD and /or end of treatment (EOT). Serial biopsies are optional for participants in Part 1a and 1c.
* Female participants must have a negative serum or urine pregnancy test within 72 hours prior to the date of the first dose of study medication if of childbearing potential or be of non-childbearing potential. Non-childbearing potential is defined as:

  * Participants >=45 years of age and has not had menses for >1 year.
  * Amenorrheic for <2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation.
  * Post hysterectomy, bilateral oophorectomy, or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
* Female participants of childbearing potential (that is [ie], those who do not meet above criteria) must agree to use 2 highly effective forms of contraception with their partners, starting with the screening visit through 150 days after the last dose of study therapy.
* The participant must have an ECOG PS of <=1.
* The participant has adequate hematologic and organ function, defined as:

  * Absolute neutrophil count (ANC) >=1500 per microliter (/μL).
  * Platelets >=100,000/μL.
  * Hemoglobin (Hb) >=9 grams per deciliter (g/dL) or >=5.6 millimoles per liter (mmol/L).
  * Serum creatinine <=1.5 times upper limit of normal (× ULN) or calculated creatinine clearance (CrCL) >=50 milliliters per minute (mL/min) using Cockcroft-Gault equation for participants with creatinine levels >1.5 × institutional ULN
  * Total bilirubin <=1.5 × ULN and direct bilirubin <=1× ULN (in the event that the total bilirubin result exceeds the upper institutional limits of normal, direct bilirubin will be obtained to determine eligibility).
  * AST and ALT <=2.5 × ULN unless liver metastases are present, in which case they must be <=5 × ULN.
  * INR of PT <=1.5 × ULN, unless participant is receiving anticoagulant therapy, then PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants; aPTT) <= 1.5 × ULN unless participant is receiving anticoagulant therapy, then PT or PTT is within therapeutic range of intended use of anticoagulants.

Inclusion criteria for participants in Part 2:

* The participant is >= 18 years of age.
* The participant has any histologically or cytologically confirmed CRC that is metastatic or not amenable to potentially curative resection (advanced), in the opinion of the Investigator.
* The participant has a primary and/or metastatic tumor(s) that is known to be MSS, as determined locally.
* The participant must have lesions amenable for biopsy and agree to undergo biopsies for fresh tumor tissue prior to treatment, approximately 4 to 6 weeks after, and, whenever possible, at EOT and/or the time of PD. If the participant has had a biopsy prior to entering the 28-day screening period, and within approximately 12 weeks of study treatment, that biopsy sample may be accepted as the Baseline fresh biopsy. Additionally, submission of sufficient high-quality archival tumor tissue is recommended, if available, to enable a longitudinal analysis of tumor biomarkers.
* The participant has measurable disease by RECIST v1.1.
* The participant has resolution to Grade <=1, per CTCAE v5.0, of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy, with the exception of peripheral neuropathy, which must have resolved to Grade <=2, and except where otherwise noted in the eligibility criteria.
* Female participants must have a negative serum or urine pregnancy test within 72 hours prior to the date of the first dose of study medication if of childbearing potential or be of non-childbearing potential. Non-childbearing potential is defined as:

  * Participants >=45 years of age and has not had menses for >1 year.
  * Amenorrheic for <2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation.
  * Post hysterectomy, bilateral oophorectomy, or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
* Female participants of childbearing potential (ie, those who do not meet above criteria) must agree to use 2 highly effective forms of contraception with their partners, starting with the screening visit through 150 days after the last dose of study therapy.
* The participant has an ECOG PS of <=1.
* The participant has adequate hematologic and organ function, defined as:

  * ANC >=1500/μL.
  * Platelets >=100,000/μL.
  * Hb >=9 g/dL or >=5.6 mmol/L.
  * Serum creatinine <=1.5 × ULN or calculated CrCL >=50 mL/min using Cockcroft-Gault equation for participants with creatinine levels >1.5 × institutional ULN
  * Total bilirubin <=1.5 × ULN and direct bilirubin <=1× ULN (in the event that the total bilirubin result exceeds the upper institutional limits of normal, direct bilirubin will be obtained to determine eligibility).
  * AST and ALT <=2.5 × ULN unless liver metastases are present, in which case they must be <=5 × ULN.
  * INR of PT <=1.5 × ULN, unless participant is receiving anticoagulant therapy, then PT or PTT is within therapeutic range of intended use of anticoagulants; aPTT) <= 1.5 × ULN unless participant is receiving anticoagulant therapy, then PT or PTT is within therapeutic range of intended use of anticoagulants.
  * Urinary protein is <=1+ on dipstick for routine urinalysis; if urine protein >=2+, a 24-hour urine sample must be collected and must demonstrate <1000 mg of protein in 24 hours to allow participation in the study.
  * Baseline albumin >=3.0 g/dL.

Inclusion Criteria for participants in Part 2A:

* The participant must have had at least 2, but no more than 3, prior lines of therapy in the advanced or metastatic setting. Adjuvant chemotherapy with radiographic progression >12 months after the last dose will not be considered a line of therapy.
* The participant has progressed on standard therapies or withdrawn from standard treatment due to unacceptable toxicity. Previous standard treatment must include all of the following:

  * Fluoropyrimidine.
  * Oxaliplatin: Participants treated with oxaliplatin in adjuvant setting should have progressed after 12 months of completion of adjuvant therapy or they must have been treated with oxaliplatin for metastatic disease.
  * Irinotecan.
  * Participants whose disease is known to be RAS-wild-type must have been treated with cetuximab, panitumumab, or other epidermal growth factor receptor (EGFR) inhibitor for metastatic disease.
  * Bevacizumab and/or another anti-angiogenic agent.
  * Previous treatment with regorafenib and/or TAS-102 are allowed in the absence of contraindications and if these agents are available to the participant according to local standards.
* The time between a participants's last chemotherapy and enrollment must be <=8 weeks.

Inclusion Criteria for participants in Part 2B:

* The participant has received <=2 prior systemic chemotherapy regimens in any setting (only 1 prior regimen for metastatic disease is permitted).

Inclusion Criteria for participants in Part 2 Cohort B1:

* The participant has received first-line combination therapy consisting of bevacizumab or anti-EGFR antibodies with FOLFIRI and has experienced radiographic progression during or after first-line therapy. Radiographic progression >12 months after the last dose of adjuvant therapy will not be considered a line of therapy.
* mFOLFOX6 therapy with bevacizumab is appropriate for the participant and is recommended by the investigator.

Inclusion Criteria for participants in Part 2 Cohort B2:

* The participant has received first-line combination therapy consisting of bevacizumab or anti-EGFR antibodies with FOLFOX (or variant) and has experienced radiographic progression during or after first-line therapy. Radiographic progression >12 months after the last dose of adjuvant therapy will not be considered a line of therapy.
* FOLFIIRI therapy with bevacizumab is appropriate for the participant and is recommended by the investigator.

Exclusion Criteria for all participants:

* The participant has previously been treated with an anti-LAG-3 antibody.
* The participant has known uncontrolled central nervous system (CNS) metastases and/or carcinomatous meningitis.
* The participant has a known concurrent, serious, uncontrolled medical disorder, nonmalignant systemic disease, or active infection requiring systemic therapy, including human immunodeficiency virus (HIV), known active hepatitis B or hepatitis C, active infection, or active autoimmune disease.
* The participant is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study.
* The participant has a history of interstitial lung disease.
* The participant has not recovered (ie, to Grade <=1 or to Baseline) from radiation- and chemotherapy-induced AEs, has received transfusion of blood products (including platelets or red blood cells), or has received administration of colony stimulating factors (including granulocyte colony-stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 3 weeks prior to the first dose of study drug.
* The participant is currently participating in an investigational study (therapy or device) or has participated in an investigational study within 4 weeks prior to the first dose of study drug.
* The participant has received prior anticancer therapy (chemotherapy, targeted therapies, radiotherapy, or immunotherapy) within 21 days or less than 5 times the half-life of the most recent therapy prior to the first dose of the drug, whichever is shorter.
* The participant has received wide-field (full-dose pelvic) radiotherapy within 28 days prior to the first dose of study drug.
* The participant has a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders.
* The participant has experienced any arterial thrombotic or arterial thromboembolic events, including, but not limited to myocardial infarction, transient ischemic attack, or cerebrovascular accident, within 12 months prior to first dose of study drug.
* The participant has received a prior autologous or allogeneic organ or transplantation.
* The participant has undergone major surgery within 28 days or subcutaneous venous access device placement within 7 days prior to the first dose of study drug.
* The participant has had a serious non-healing wound, ulcer, or bone fracture within 28 days prior to first dose of study drug.
* The participant has an elective or planned major surgery to be performed during the course of the trial.
* The participant has a history of inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) in the 12 months prior to the first dose of study drug.
* The participant has an acute or subacute bowel obstruction, abdominal fistula, or history of chronic diarrhea which is considered clinically significant, in the opinion of the investigator.
* The participant has experienced a Grade >=3 bleeding event within 3 months prior to the first dose of study drug.
* The participant has either peptic ulcer disease associated with a bleeding event or known active diverticulitis.
* The participant has not recovered (Grade >=1) from AEs and/or complications from any major surgery prior to the first dose of study drug.
* The participant has received a vaccine within 7 days of the first dose of study drug.
* The participant has known hypersensitivity to TSR-033, dostarlimab (Part 1c and Part 2), or associated excipients.

Exclusion Criteria for participants in Part 1:

* The participant's prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-LAG-3 agent that resulted in permanent discontinuation due to an AE.

Exclusion Criteria for participants in Part 2:

* The participant has been previously treated with an anti-PD-1 or anti-PD-L1 antibody.

Exclusion Criteria for participants in Part 2B:

* The participant has known dihydropyrimidine dehydrogenase deficiency.
* The participant experienced an arterial thrombotic/thromboembolic event, Grade 4 hypertension, Grade 4 proteinuria, a Grade 3-4 bleeding event, or bowel perforation during first-line therapy with a bevacizumab-containing regimen.
* The participant has known hypersensitivity to bevacizumab, mFOLFOLX6 (Cohort B1) or FOLFIRI (Cohort B2), or associated excipients.
* The participant experienced PD within 12 months of last dose of adjuvant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2023-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (11):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hecht JR, Michot JM, Bajor D, Patnaik A, Chung KY, Wang J, Falchook G, Cleary JM, Kim R, Krishnamurthy A, Marathe O, Youssoufian H, Ellis C, Waszak A, Ghosh S, Zhang H, Yablonski K, Shah SD, Diaz-Padilla I, Ulahannan S. CITRINO: phase 1 dose escalation study of anti-LAG-3 antibody encelimab alone or in combination with anti-PD-1 dostarlimab in patients with advanced/metastatic solid tumours. BJC Rep. 2025 Feb 27;3(1):10. doi: 10.1038/s44276-024-00118-x. PMID 40016550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was comprised of two parts. Part 1 was a dose escalation phase and consisted of two cohorts 1AB and 1C. Part 2 was Colorectal Cancer dose expansion phase and consisted of 3 cohorts 2A, 2B1 and 2B2.
Groups:
- Part 1AB - TSR-033 [20 Milligrams (mg)]: In part 1a, participants with advanced or metastatic solid tumors received 20 mg TSR-033 via 30-minute intravenous (IV) infusion once every 2 weeks (Q2W).
- Part 1AB - TSR-033 (80 mg): In part 1a, participants with advanced or metastatic solid tumors received 80 mg TSR-033 via 30-minute IV infusion once Q2W. In part 1b, additional participants enrolled in this dose level to characterize the PK profile of TSR-033 and assess PDy data followed by treatment with TSR-033 dosed on day 1, and then once Q2W.
- Part 1AB - TSR-033 (240 mg): In part 1a, participants with advanced or metastatic solid tumors received 240 mg TSR-033 via 30-minute IV infusion once Q2W. In part 1b, additional participants enrolled in this dose level to characterize the PK profile of TSR-033 and assess PDy data followed by treatment with TSR-033 dosed on day 1, and then once Q2W.
- Part 1AB - TSR-033 (720 mg): In part 1a, participants with advanced or metastatic solid tumors received 720 mg TSR-033 via 30-minute IV infusion once Q2W. In part 1b, additional participants enrolled in this dose level to characterize the PK profile of TSR-033 and assess PDy data followed by treatment with TSR-033 dosed on day 1, and then once Q2W.
- Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg): Participants with advanced or metastatic solid tumors received 80 mg TSR-033 via 30-minute IV infusion in combination with 500 mg dostarlimab on day 1, and then once every 3 weeks (Q3W).
- Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg): Participants with advanced or metastatic solid tumors received 240 mg TSR-033 via 30-minute IV infusion in combination with 500 mg dostarlimab on day 1, and then once Q3W.
- Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg): Participants with advanced or metastatic solid tumors received 720 mg TSR-033 via 30-minute IV infusion in combination with 500 mg dostarlimab on day 1, and then once Q3W.
- Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg); PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg): Anti-programmed cell death-1 receptor (PD-1) naive participants with advanced or metastatic microsatellite stable colorectal cancer (MSS-CRC) that progressed following 2 or 3 prior lines of therapy received IV infusion of 720 mg TSR-033 once Q2W in combination with 1000 mg dostarlimab once every 6 weeks (Q6W).
- Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6: Anti-PD-1-naive participants with advanced or metastatic MSS-CRC following progression on frontline treatment with FOLFIRI (or variant), with or without biologics received IV infusion of 720 mg TSR-033 once (on day 3 of each cycle) Q2W in combination with 1000 mg dostarlimab once (on day 3 of each cycle) Q6W and mFOLFOX6 (on day 1 of each cycle) Q6W and 30-minute IV infusion of bevacizumab (bev) once (on day 1 of each cycle) Q6W. As a part of mFOLFOX6 regimen combination of 2-hour infusion of oxaliplatin with leucovorin and 2-4 minutes infusion of 5-Fluorouracil on day 1 along with continuous 46-hours infusion of 5-Fluorouracil on day 1 to day 3 were administered.
- Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI; PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI: Anti-PD-1-naive participants with advanced or metastatic MSS-CRC following progression on frontline treatment with FOLFOX (or variant), with or without biologics received IV infusion of 720 mg TSR-033 once (on day 3 of each cycle) Q2W in combination with 1000 mg dostarlimab once (on day 3 of each cycle) Q6W and FOLFIRI (on day 1 of each cycle) Q6W and 30-minute IV infusion of bevacizumab (bev) once (on day 1 of each cycle) Q6W. As a part of FOLFIRI regimen combination of 90 minutes infusion of Irinotecan with leucovorin with 2-4 minutes infusion of 5-Fluorouracil on day 1 and continuous 46-hours infusion of 5-Fluorouracil on day 1 to day 3 were administered.
Period: Part 1 (Up to Approximately 51 Months)
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg) | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg) | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Started | 3 | 10 | 11 | 10 | 5 | 7 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 10 | 11 | 10 | 5 | 7 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 6 | 5 | 5 | 3 | 6 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 5 | 5 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2A (Up to Approximately 30 Months)
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg) | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg) | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 2B (Up to Approximately 29 Months)
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg) | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg) | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (New participants started and dosed in this part.) | 21 (New participants started and dosed in this part.) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 20 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 0
Period: PACT Phase (up to Approximately 36weeks)
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg) | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg) | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (Participant completing the Period 2A entered into PACT Phase) | 1 (Participant completing the treatment plan under the 2B2 entered into PACT phase.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg) | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg) | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI | Total
Number analyzed (Participants) | 3 | 10 | 11 | 10 | 5 | 7 | 6 | 34 | 4 | 21 | 111
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  19 - 64 years | 1 | 5 | 6 | 6 | 4 | 4 | 5 | 25 | 3 | 17 | 76
  >=65 years | 2 | 5 | 5 | 4 | 1 | 3 | 1 | 9 | 1 | 4 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 5 | 4 | 2 | 3 | 5 | 18 | 0 | 5 | 51
  Male | 1 | 3 | 6 | 6 | 3 | 4 | 1 | 16 | 4 | 16 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 8 | 7 | 7 | 3 | 4 | 5 | 28 | 3 | 15 | 83
  Black | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 3 | 9
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 4
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
  Other | 0 | 1 | 4 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 12

OUTCOME MEASURES:

1. Secondary Outcome: Part 1ab: Area Under the Concentration-time Curve From Time Zero to Last Measurable Concentration (AUC [0-last]) of TSR-033
Description: Blood samples were collected for pharmacokinetic (PK) analysis of TSR-033 when administered intravenously as monotherapy. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1.5, 3, 24, 48, 96 and 168 hour
Population: Pharmacokinetic (PK) population included all partiocipants who received any amount of TSR 033 and/or dostarlimab and have ≥1 measurable drug concentration. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram/millilitre (h*ug/mL)
Groups:
- Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg): In part 1a, participants with advanced or metastatic solid tumors received 720 mg TSR-033 via 30-minute IV infusion once Q2W. In part 1b, additional participants enrolled in this dose level to characterize the PK profile of TSR-033 and assess PDy data followed by treatment with TSR-033 dosed on day 1, and then once Q2W.
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 3 | 10 | 10 | 10
Hour*microgram/millilitre (h*ug/mL) | 606.4256 (32.65) | 2601.731 (70.3423) | 8176.4963 (29.4644) | 23763.7645 (48.7606)

2. Secondary Outcome: Part 1c: AUC (0-last) of TSR-033 and Dostarlimab
Description: Blood samples were collected for PK analysis of TSR-033 when administered intravenously in combination with dostarlimab. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1, 1.5, 3, 24, 48, 96, 168, 336 and 504 hour
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 7 | 6
h*ug/mL
  TSR-033 | 2615.4485 (33.8335) | 9317.8306 (21.9902) | 30750.7484 (28.6869)
  Dostarlimab | 24303.8328 (31.4148) | 25301.7468 (17.9326) | 26326.0589 (26.9526)

3. Secondary Outcome: Part 1ab: AUC Extrapolated From Time Zero to Infinity (AUC [0-inf]) of TSR-033
Description: Blood samples were collected for PK analysis of TSR-033 when administered intravenously as monotherapy. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1.5, 3, 24, 48, 96 and 168 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 2 | 3 | 5 | 5
h*ug/mL | 858.3739 (39.3306) | 2783.4404 (112.7081) | 12517.0356 (37.2816) | 44300.8914 (32.4781)

4. Secondary Outcome: Part 1c: AUC (0-inf) of TSR-033 and Dostarlimab
Description: as for outcome 2
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1, 1.5, 3, 24, 48, 96, 168, 336 and 504 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 4 | 3
h*ug/mL
  TSR-033 | 3201.6715 (35.5887) | 12336.2784 (26.1779) | 52144.2561 (15.6182)
  Dostarlimab: number analyzed (Participants) | 2 | 1 | 2
  Dostarlimab | 30692.5087 (26.1453) | 34298.0046 (NA) — Geometric coefficient of variation is not applicable as only a single participant was analyzed. | 37944.78 (25.3851)

5. Secondary Outcome: Part 1ab: AUC Over a Dosing Interval at Steady State (AUCtau) of TSR-033
Description: as for outcome 3
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1.5, 3, 24, 48, 96 and 168 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 3 | 8 | 10 | 8
h*ug/mL | 816.9529 (32.427) | 3171.9548 (52.272) | 9432.5708 (23.5407) | 27125.0835 (27.0846)

6. Secondary Outcome: Part 1c: AUCtau of TSR-033 and Dostarlimab
Description: as for outcome 2
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1, 1.5, 3, 24, 48, 96, 168, 336 and 504 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 7 | 5
h*ug/mL
  TSR-033: number analyzed (Participants) | 5 | 6 | 5
  TSR-033 | 2929.7274 (34.6086) | 11351.945 (26.8461) | 39920.9217 (19.2402)
  Dostarlimab | 29866.3126 (33.313) | 32396.6385 (19.5917) | 32702.9638 (31.1208)

7. Secondary Outcome: Part 1ab: Maximum Concentration (Cmax) of TSR-033
Description: as for outcome 3
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1.5, 3, 24, 48, 96 and 168 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 3 | 10 | 10 | 10
ug/mL | 7.489 (30.807) | 22.81 (29.88) | 74.13 (21.35) | 217.1 (34.8)

8. Secondary Outcome: Part 1c: Cmax of TSR-033 and Dostarlimab
Description: as for outcome 2
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1, 1.5, 3, 24, 48, 96, 168, 336 and 504 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 7 | 6
ug/mL
  TSR-033 | 23.04 (29.09) | 73.5 (13.8) | 312.8 (79.4)
  Dostarlimab | 171.6 (34.5) | 163 (17.2) | 170.8 (27)

9. Secondary Outcome: Part 1ab: Clearance (CL) of TSR-033
Description: as for outcome 3
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1.5, 3, 24, 48, 96 and 168 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre/ hour (L/h)
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 2 | 3 | 5 | 5
Litre/ hour (L/h) | 0.0233 (39.3306) | 0.0287 (112.7081) | 0.0192 (37.2816) | 0.0163 (32.4781)

10. Secondary Outcome: Part 1c: CL of TSR-033 and Dostarlimab
Description: as for outcome 2
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1, 1.5, 3, 24, 48, 96, 168, 336 and 504 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 4 | 3
L/h
  TSR-033 | 0.025 (35.5887) | 0.0195 (26.1779) | 0.0138 (15.6182)
  Dostarlimab: number analyzed (Participants) | 2 | 1 | 2
  Dostarlimab | 0.0163 (26.1453) | 0.0146 (NA) — Geometric coefficient of variation is not applicable as only a single participant was analyzed. | 0.0132 (25.3851)

11. Secondary Outcome: Part 1ab: Volume of Distribution at Steady State (Vss) of TSR-033
Description: as for outcome 3
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1.5, 3, 24, 48, 96 and 168 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 3 | 8 | 10 | 8
Litre | 3.4821 (36.6086) | 5.0563 (33.1027) | 4.8329 (21.6021) | 5.2564 (31.2434)

12. Secondary Outcome: Part 1c: Vss of TSR-033 and Dostarlimab
Description: as for outcome 2
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1, 1.5, 3, 24, 48, 96, 168, 336 and 504 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 7 | 5
Litre
  TSR-033: number analyzed (Participants) | 5 | 6 | 5
  TSR-033 | 4.8162 (36.8613) | 5.3978 (17.3282) | 4.3845 (32.7955)
  Dostarlimab | 4.4915 (36.0302) | 4.6431 (13.0127) | 4.3544 (34.1792)

13. Secondary Outcome: Part 1ab: Terminal Half-life (t1/2) of TSR-033
Description: as for outcome 3
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1.5, 3, 24, 48, 96 and 168 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 3 | 8 | 10 | 8
Hour | 119.7937 (19.1377) | 240.5387 (72.7919) | 198.8801 (39.3322) | 214.2533 (32.6387)

14. Secondary Outcome: Part 1c: t1/2 of TSR-033 and Dostarlimab
Description: as for outcome 2
Time Frame: Pre-dose and post-dose 15 minute, 30 minute, 1, 1.5, 3, 24, 48, 96, 168, 336 and 504 hour
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 7 | 5
Hour
  TSR-033: number analyzed (Participants) | 5 | 6 | 5
  TSR-033 | 140.4589 (18.3381) | 241.0348 (25.7829) | 226.5019 (26.7142)
  Dostarlimab | 259.3884 (33.9148) | 318.7548 (18.7546) | 286.253 (23.726)

15. Secondary Outcome: Part 1ab: Number of Participants With Anti-TSR-033 Antibodies
Description: Serum samples will be collected and tested for the presence of antibodies to TSR-033.
Time Frame: Up to 51 months
Population: Immunogenicity (ADA) population included all participants who received at least 1 dose of TSR-033 and who have at least 1 ADA sample with a result. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 3 | 10 | 11 | 9
Participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Part 1c: Number of Participants With Anti-TSR-033 Antibodies
Description: Serum samples will be collected and tested for the presence of antibodies to TSR-033.
Time Frame: Up to 29 months
Population: Immunogenicity (ADA) population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 7 | 6
Participants | 1 | 0 | 0

17. Secondary Outcome: Part 2A: Number of Participants With Anti-TSR-033 Antibodies
Description: Serum samples will be collected and tested for the presence of antibodies to TSR-033.
Time Frame: Up to 29 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg)
Number analyzed (Participants) | 21
Participants | 0

18. Secondary Outcome: Part 2B: Number of Participants With Anti-TSR-033 Antibodies
Description: Serum samples will be collected and tested for the presence of antibodies to TSR-033.
Time Frame: Up to 29 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 20
Participants | 0 | 0

19. Secondary Outcome: Part 1ab: Objective Response Rate (ORR)
Description: ORR is defined as percentage of participants achieving complete response (CR) or partial response (PR) as assessed by the investigator per response evaluation criteria in solid tumors (RECIST)v1.1. CR defined as disappearance of all target & non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 51 months
Population: Efficacy population included all participants who received any amount of TSR-033.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB: TSR-033:Part 1AB - TSR-033 (720 mg)
Number analyzed (Participants) | 3 | 10 | 11 | 10
Percentage of participants | 0 [0 to 70.8] | 0 [0 to 30.8] | 0 [0 to 28.5] | 0 [0 to 30.8]

20. Secondary Outcome: Part 1c: Objective Response Rate (ORR)
Description: as for outcome 19
Time Frame: Up to 29 months
Population: Efficacy population included all participants who received any amount of TSR-033.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 7 | 6
Percentage of participants | 0 [0 to 52.2] | 0 [0 to 41] | 0 [0 to 45.9]

21. Secondary Outcome: Part 2B: Objective Response Rate (ORR)
Description: as for outcome 19
Time Frame: Up to 29 months
Population: Efficacy population included all participants who received any amount of TSR-033.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 20
Percentage of participants | 0 [0 to 60.2] | 20 [5.7 to 43.7]

22. Secondary Outcome: Part 2A: Duration of Response (DOR)
Description: DOR was defined as the time from first documentation of CR or PR by RECIST v1.1 until the time offirst documentation of PD per RECIST v1.1. CR defined as disappearance of all target & non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 29 months
Population: Efficacy population. Only responders by investigator assessment were included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg)
Number analyzed (Participants) | 1
Months | 23.3 [23.3 to 23.3]

23. Secondary Outcome: Part 2B: Duration of Response (DOR)
Description: as for outcome 22
Time Frame: Up to 29 months
Population: Efficacy population. Only responders by investigator assessment were included in this analysis. There were no responders in the arm Part 2B1, hence the participants analysed in 0.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 0 | 4
Months |  | 14.1 [6.7 to 19.2]

24. Secondary Outcome: Part 2A: Disease Control Rate (DCR)
Description: DCR is defined as defined as the percentage of participants achieving CR, PR, or stable disease (SD) as assessedby the investigator per RECIST v1.1. CR defined as disappearance of all target & non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
Time Frame: Up to 29 months
Population: Efficacy population. Only responders by investigator assessment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg)
Number analyzed (Participants) | 34
Percentage of participants | 8.8 [1.9 to 23.7]

25. Secondary Outcome: Part 2B: Disease Control Rate (DCR)
Description: as for outcome 24
Time Frame: Up to 29 months
Population: Efficacy population. Only responders by investigator assessment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 20
Percentage of participants | 50 [6.8 to 93.2] | 80 [56.3 to 94.3]

26. Primary Outcome: Part 1A: Number of Participants Experiencing Dose Limiting Toxicity (DLT)
Description: DLTs were assessed based on common terminology criteria for adverse events (CTCAE) v5.0 included drug-related AEs like grade>=2 uveitis, eye pain, or blurred vision that does not resolve with topical therapy within 2 weeks, grade ≥2 immune-related endocrine toxicity that required hormone replacement, grade 2 or 3 colitis or diarrhea that persisted without resolution to grade<=1 for >=7days despite adequate immune suppressive therapy, grade 3 or 4 immune-related AEs (irAE) without resolution to grade<=1 or baseline within 8 days despite adequate immune suppressive therapy, any grade clinically significant (CS) irAE requiring treatment discontinuation, other grade>=3 non-hematologic toxicity, any CS grade>=3 non-hematologic laboratory abnormality, any CS hematologic toxicity and any death that is not clearly attributed to the underlying disease or extraneous causes. CTCAE defines Grade 0 as normal, 1 as mild, 2 as moderate, 3 as severe and Grade 4 as life-threatening consequences.
Time Frame: Up to 28 days
Population: DLT evaluable population included only those participants who completed the DLT observation period throughout the course of 2 TSR-033 administrations (Day 1 and Day 15 in the first 28 days of study treatment) for Part 1A unless the participant discontinued TSR-033 (Part 1A) due to a DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1A - TSR-033 [20 Milligrams (mg)]: In part 1A, participants with advanced or metastatic solid tumors received 20 mg TSR-033 via 30-minute intravenous (IV) infusion once every 2 weeks (Q2W).
- Part 1A - TSR-033 (80 mg): In part 1A, participants with advanced or metastatic solid tumors received 80 mg TSR-033 via 30-minute IV infusion once Q2W.
- Part 1A - TSR-033 (240 mg): In part 1A, participants with advanced or metastatic solid tumors received 240 mg TSR-033 via 30-minute IV infusion once Q2W.
- Part 1A - TSR-033 (720 mg): In part 1A, participants with advanced or metastatic solid tumors received 720 mg TSR-033 via 30-minute IV infusion once Q2W.
Arm/Group | Part 1A - TSR-033 [20 Milligrams (mg)] | Part 1A - TSR-033 (80 mg) | Part 1A - TSR-033 (240 mg) | Part 1A - TSR-033 (720 mg)
Number analyzed (Participants) | 3 | 6 | 6 | 6
Participants | 0 | 1 | 0 | 0

27. Primary Outcome: Part 1C: Number of Participants Experiencing DLT
Description: as for outcome 26
Time Frame: Up to 42 days
Population: DLT evaluable population included the assessment of DLTs in Part 1C included only those participants who completed the DLT observation period throughout the course of 2 TSR-033 + dostarlimab administrations (Day 1 and Day 21 in the first 42 days of study treatment), for Part 1C unless the participant discontinued TSR-033 + dostarlimab (Part 1C) due to a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 5 | 7 | 6
Participants | 0 | 0 | 0

28. Primary Outcome: Part 2B: Number of Participants Experiencing DLT
Description: as for outcome 26
Time Frame: Up to 30 days
Population: DLT evaluable population included the assessment of DLTs in Part 2B included only those participants completing the DLT observation period throughout the course of 2 TSR-033 + dostarlimab administrations (Day 3 and Day 17 in the first 30 days of study treatment), for Part 2B unless the participant discontinued TSR-033 + dostarlimab (Part 2B) due to a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 21
Participants | 0 | 0

29. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs), Treatment-emergent AEs (TEAEs)and Immune-related AEs (irAEs)
Description: SAEs are any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. TEAEs are defined as any new AE that begins, or any pre-existing condition that worsens in severity, after at least 1 dose of study treatment administration. Immune-related adverse events of interest (irAEs) are defined as any >= Grade 2 AEs based on a pre-specified list. CTCAE defines Grade 0 as normal, 1 as mild, 2 as moderate, 3 as severe and Grade 4 as life-threatening consequences.
Time Frame: Up to approximately 51 months
Population: Safety population included all participants who receive any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 3 | 10 | 11 | 10 | 5 | 7 | 6
Participants
  SAEs | 1 | 5 | 2 | 1 | 1 | 3 | 4
  TEAEs | 3 | 10 | 10 | 10 | 5 | 7 | 6
  irAEs | 0 | 4 | 2 | 2 | 2 | 3 | 4

30. Primary Outcome: Part 2B: Number of Participants With SAEs, TEAEs and irAEs
Description: as for outcome 29
Time Frame: Up to approximately 29 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 21
Participants
  SAEs | 4 | 7
  TEAEs | 4 | 21
  irAEs | 3 | 11

31. Primary Outcome: Part 1: Number of Participants With Grade Shift From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters and each parameter was graded according to national cancer institute (NCI)-common terminology criteria for adverse events (CTCAE) version 5.0. Grade 0: normal, Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent non-missing measurement prior to the first administration of study drug. Data has been presented for the number of participants with hematology grade shifts from baseline grade to grade 3 and 4 for each parameter.
Time Frame: Up to 51 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 3 | 10 | 11 | 10 | 5 | 7 | 6
Participants
  Hemoglobin, Grade 1 to Grade 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Hemoglobin, Grade 2 to Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Grade 0 to Grade 3 | 0 | 2 | 0 | 0 | 1 | 1 | 1
  Lymphocytes, Grade 2 to Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Lymphocytes, Grade 3 to Grade 3 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  Neutrophils, Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1

32. Primary Outcome: Part 2B: Number of Participants With Grade Shift From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters and each parameter was graded according to national cancer institute (NCI)-common terminology criteria for adverse events (CTCAE) version 5.0. Grade 0: normal, Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent non-missing measurement prior to the first administration of study drug. Data have been presented for the number of participants with hematology grade shifts from baseline grade to grade 3 and 4 for each parameter. WBC is white blood cells.
Time Frame: Up to 29 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 21
Participants
  Hemoglobin, Grade 2 to Grade 3 | 0 | 2
  Lymphocytes, Grade 0 to Grade 3 | 1 | 2
  Lymphocytes, Grade 0 to Grade 4 | 1 | 0
  Lymphocytes, Grade 2 to Grade 3 | 0 | 4
  Neutrophils, Grade 0 to Grade 3 | 1 | 8
  Neutrophils, Grade 0 to Grade 4 | 1 | 1
  Platelets, Grade 0 to Grade 3 | 0 | 1
  WBC (Leukopenia), Grade 0 to Grade 3 | 1 | 4
  WBC (Leukopenia), Grade 0 to Grade 4 | 1 | 0

33. Primary Outcome: Part 1: Number of Participants With Grade Shift From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of clinical chemistry parameters and each parameter was graded according to national cancer institute (NCI)-common terminology criteria for adverse events (CTCAE) version 5.0. Grade 0: normal, Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent non-missing measurement prior to the first administration of study drug. Data have been presented for the number of participants with clinical chemistry grade shifts from baseline grade to grade 3 and 4 for each parameter.
Time Frame: Up to 51 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 3 | 10 | 11 | 10 | 5 | 7 | 6
Participants
  Hyperkalemia, Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypoalbuminemia, Grade 2 to Grade 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Hypokalemia, Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypomagnesemia, Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1

34. Primary Outcome: Part 2B: Number of Participants With Grade Shift From Baseline in Clinical Chemistry Parameters
Description: as for outcome 33
Time Frame: Up to 29 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 21
Participants
  Hypercalcemia, Grade 0 to Grade 4 | 0 | 2
  Hypocalcemia, Grade 0 to Grade 4 | 0 | 2

35. Primary Outcome: Part 1: Number of Participants With Grade 3 and 4 Toxicities in Clinical Chemistry Parameters - Creatinine, Bilirubin, Alkaline Phosphatase
Description: Blood samples were collected for the analysis of clinical chemistry parameters and each parameter was graded according to national cancer institute (NCI)-common terminology criteria for adverse events (CTCAE) version 5.0. Grade 0: normal, Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Data have been presented for the number of participants with clinical chemistry grade3 and 4 toxicities each parameter.
Time Frame: Up to 51 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 3 | 10 | 11 | 10 | 5 | 7 | 6
Participants
  Alkaline phosphatase | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bilirubin | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Creatinine | 0 | 0 | 0 | 0 | 0 | 0 | 1

36. Primary Outcome: Part 2B: Number of Participants With Grade 3 and 4 Toxicities in Clinical Chemistry Parameters - Alanine Aminotransferase, Aspartate Aminotransferase, Creatinine, Bilirubin
Description: Blood samples were collected for the analysis of clinical chemistry parameters and each parameter was graded according to national cancer institute (NCI)-common terminology criteria for adverse events (CTCAE) version 5.0. Grade 0: normal, Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the most recent non-missing measurement prior to the first administration of study drug. Data have been presented for the number of participants with clinical chemistry grade 3 and 4 toxicities each parameter.
Time Frame: Up to 29 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 21
Participants
  Alanine aminotransferase | 1 | 0
  Aspartate aminotransferase | 1 | 1
  Bilirubin | 1 | 2
  Creatinine | 0 | 1

37. Primary Outcome: Part 1: Number of Participants With Post Baseline Abnormal Electrocardiogram (ECG) Results
Description: 12-lead ECG were obtained using an ECG machine. Participants were in supine or a semi-recumbent position (about 30 degrees of elevation) and rested for approximately 2 minutes before ECGs are recorded. ECG results included QT interval corrected for heart rate according to Bazett's formula (QTcB), QT interval corrected for heart rate according to Fridericia's formula (QTcF), QRS interval, PR Interval and Heart rate.
Time Frame: Up to 51 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg)
Number analyzed (Participants) | 3 | 10 | 11 | 10 | 5 | 7 | 6
Participants
  QTcF | 1 | 2 | 1 | 0 | 0 | 0 | 0
  QTcB | 1 | 1 | 0 | 0 | 0 | 1 | 1
  QRS | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Heart Rate | 0 | 0 | 0 | 0 | 1 | 1 | 0
  PR Interval | 0 | 0 | 1 | 0 | 0 | 0 | 0

38. Primary Outcome: Part 2B: Number of Participants With Post Baseline Abnormal ECG Results
Description: as for outcome 37
Time Frame: Up to 29 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
Number analyzed (Participants) | 4 | 21
Participants
  QTcF | 1 | 2
  QTcB | 1 | 5
  QRS | 1 | 2
  Heart Rate | 0 | 2
  PR Interval | 0 | 1

39. Primary Outcome: Part 2A: Objective Response Rate (ORR)
Description: ORR is defined as percentage of participants achieving complete response (CR) or partial response (PR) as assessed by the investigator per response evaluation criteria in solid tumors (RECIST)v1.1. CR defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 30 months
Population: Efficacy population included all participants who received any amount of TSR-033.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg)
Number analyzed (Participants) | 34
Percentage of participants | 2.9 [0.1 to 15.3]

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected maximum up to 51 months for Part 1 and up to approximately 29 months for Part 2A and up to 29 months for Part 2B and and from month 51 to week 36 for PACT phase.
Description: Safety population included all participants who receive any amount of any study drug.
Arm/Group | Part 1AB - TSR-033 [20 Milligrams (mg)] | Part 1AB - TSR-033 (80 mg) | Part 1AB - TSR-033 (240 mg) | Part 1AB - TSR-033 (720 mg) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg) | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg) | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI
All-Cause Mortality (participants affected / at risk) | 1/3 | 6/10 | 5/11 | 5/10 | 3/5 | 6/7 | 3/6 | 18/34 | 1/4 | 7/21 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 5/10 | 2/11 | 1/10 | 1/5 | 3/7 | 4/6 | 8/34 | 4/4 | 7/21 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10 | 11/11 | 10/10 | 5/5 | 7/7 | 6/6 | 31/34 | 4/4 | 21/21 | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1AB - TSR-033 [20 Milligrams (mg)] (N=3) | Part 1AB - TSR-033 (80 mg) (N=10) | Part 1AB - TSR-033 (240 mg) (N=11) | Part 1AB - TSR-033 (720 mg) (N=10) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) (N=5) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) (N=7) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg) (N=6) | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg) (N=34) | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 (N=4) | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI (N=21) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) (N=1) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1AB - TSR-033 [20 Milligrams (mg)] (N=3) | Part 1AB - TSR-033 (80 mg) (N=10) | Part 1AB - TSR-033 (240 mg) (N=11) | Part 1AB - TSR-033 (720 mg) (N=10) | Part 1C - TSR-033 (80 mg) + Dostarlimab (500 mg) (N=5) | Part 1C - TSR-033 (240 mg) + Dostarlimab (500 mg) (N=7) | Part 1C - TSR-033 (720 mg) + Dostarlimab (500 mg) (N=6) | Part 2A - TSR-033 (720 mg) + Dostarlimab (1000 mg) (N=34) | Part 2B1 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev + mFOLFOX6 (N=4) | Part 2B2 - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI (N=21) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) (N=1) | PACT Phase - TSR-033 (720 mg) + Dostarlimab (1000 mg) + Bev +FOLFIRI (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 7 (12) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (5) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (5) | 1 (1) | 6 (8) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 8 (8) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 3 (7) | 10 (14) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (7) | 7 (8) | 2 (5) | 11 (13) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 2 (4) | 5 (7) | 2 (5) | 5 (7) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 3 (7) | 10 (11) | 3 (3) | 10 (18) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (3) | 5 (6) | 1 (2) | 3 (3) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 2 (4) | 10 (14) | 1 (1) | 5 (7) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (7) | 3 (4) | 1 (2) | 2 (8) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (10) | 4 (6) | 1 (1) | 2 (6) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 3 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 7 (18) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (2) | 2 (3) | 1 (1) | 1 (1) | 4 (5) | 6 (6) | 1 (1) | 4 (7) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 4 (5) | 0 (0) | 4 (9) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (5) | 1 (1) | 2 (3) | 2 (5) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (5) | 2 (3) | 2 (4) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (6) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anticipatory anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 3 (4) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (7) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 4 (11) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT03250832/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT03250832/SAP_001.pdf